CLINICAL TRIAL: NCT02270307
Title: Allogeneic Bone Marrow Transplantation (Allo-BMT) From Human Leukocyte Antigen (HLA) - Identical Related and Unrelated Donors in Patients With Hematological Malignancies With High Risk of Relapse Using Cyclophosphamide (CY) and Mesenchymal Stromal Cells (MSC) as aGVHD Prophylaxis
Brief Title: MSC and Cyclophosphamide for Acute Graft-Versus-Host Disease (aGVHD) Prophylaxis
Acronym: MSC-CY
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, PI, National Research Center for Hematology, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MSC-CY-Russia
Record Dates: First submitted 2014-04-07; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Multiple Myeloma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSC+CY (Experimental): Cyclophosphamide 50 mg/kg/day at +3, +4 day once daily after BMT Mesenchymal stromal cells 1*10^6/kg at day of recovery
  Interventions: Drug: Cyclophosphamide; Biological: Mesenchymal stromal cells

INTERVENTIONS:
Drug: Cyclophosphamide — Dose 50 mg/kg at day +3,+4 once daily
Biological: Mesenchymal stromal cells — Dose 1 million per kg, at day of recovery once

SUMMARY:
Evaluating the effectiveness of the new protocol which replace the standard immunosuppressive therapy with use of MSCs and CY in patients at high risk of relapse.

DETAILED DESCRIPTION:
This trial try to find a new way of refractory hematological malignancies treatment. Aim of this study evaluating the effectiveness of the new protocol which replace the standard immunosuppressive therapy with use of MSCs and CY in patients at high risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Refractory forms of acute leukemia, but in complete remission (CR)
* Second and third remission of acute leukemia
* 2nd and 3rd chronic phase chronic myelogenous leukemia (CML) (or Ph + ALL)
* relapsed multiple myeloma
* advanced leukemia

Exclusion Criteria:

* ICU
* Mechanical ventilation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Valery Savchenko, Prof., Study Director — Ministry of Health
Locations (1):
- BMT department, Moscow, Russia